CLINICAL TRIAL: NCT05721053
Title: Improving Outcomes for Older Adults Undergoing Radiation Therapy: Prospective Cohort Study
Brief Title: Improving Outcomes for Older Adults Undergoing Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kavita Dharmarajan, Associate Professor of Radiation Oncology, Geriatrics, and Palliative Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 19-2371; 1K76AG068516-01A1 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Radiation Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older Adults in Radiation Therapy: Older Adults who are receiving Radiation Therapy.

SUMMARY:
The purpose of this study is to improve healthcare received by people ≥ 65 years who are receiving radiation therapy (RT). The study will primarily examine patients ability to complete RT, changes in a patients' daily function and self-reported toxicities. To collect this information, study participants will be asked to complete surveys and physical and cognitive function assessments at five different timepoints in their treatment: before RT, End of RT, and at 1, 3, and 6 months follow up visits. Findings of this study will help radiation oncologists make more informed decisions for future patients receiving RT.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 65 years
* Patient must have pathologically confirmed cancer
* Patient must have the ability to provide informed consent, or have a legally authorized representative (LAR) present to provide informed consent on the participant's behalf
* Must be radiation oncology patient at Mount Sinai Hospital, Mount Sinai Downtown, or Mount Sinai West.

Exclusion Criteria:

* There is no exclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All participants presenting to Mount Sinai Hospital, Mount Sinai Downtown, and Mount Sinai West who meet eligibility criteria will be given the option of participating. The hospitals serve distinct regions of New York City with diverse sociodemographic characteristics. All have RT services for ambulatory and hospitalized patients.
  The total number of study enrollments at Mount Sinai Hospital, Mount Sinai Downtown, and Mount Sinai West twill be approximately 225 over 36 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Completion of Radiation Treatment | at end of RT, average of 10 days
  The number of patients who have completed their radiation therapy (RT).
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-30) Score Pre-RT | pre-RT, time 0
  EORTC-QLQ-30 Score consists of 30 items covered by 1 of 3 dimensions:
  * Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  * Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  * Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores are calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
EORTC-QLQ-30 Score at Post-RT | at end of RT, average of 10 days
  EORTC-QLQ-30 Score consists of 30 items covered by 1 of 3 dimensions:
  * Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  * Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  * Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores are calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
EORTC-QLQ-30 Score at 1 month follow-up | at 1 month follow-up
  EORTC-QLQ-30 Score at 1 month follow up. EORTC-QLQ-30 Score consists of 30 items covered by 1 of 3 dimensions:
  * Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  * Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  * Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores are calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
EORTC-QLQ-30 Score at 3 months follow up | at 3 months follow-up
  EORTC-QLQ-30 Score at 3 months follow up. EORTC-QLQ-30 Score consists of 30 items covered by 1 of 3 dimensions:
  * Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  * Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  * Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores are calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
EORTC-QLQ-30 Score at 6 months follow up | at 6 months follow-up
  EORTC-QLQ-30 Score at 6 months follow up. EORTC-QLQ-30 Score consists of 30 items covered by 1 of 3 dimensions:
  * Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  * Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much).
  * Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  All domain scores are calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.

SECONDARY OUTCOMES:
Short Physical Performance Battery Score at Pre-RT | pre-RT, time 0
  Physical performance pre-RT, measured by the Short Physical Performance Battery (SPPB), a 10-minute provider-administered test of balance, 4-meter walk, and chair stands, which predicts disability and mortality in older adults and cancer patients. Each of the 3 tests are scored from 0-4 and summed for a total scale range of 0-12, with higher scores indicating better physical function.
Short Physical Performance Battery Score at at 1 month follow-up | at 1 month follow-up
  Physical performance at 1 month follow-up, measured by the Short Physical Performance Battery (SPPB), a 10-minute provider-administered test of balance, 4-meter walk, and chair stands, which predicts disability and mortality in older adults and cancer patients. Each of the 3 tests are scored from 0-4 and summed for a total scale range of 0-12, with higher scores indicating better physical function.
Short Physical Performance Battery Score at 3 months follow-up | at 3 months follow-up
  Physical performance at 3 month follow-up, measured by the Short Physical Performance Battery (SPPB), a 10-minute provider-administered test of balance, 4-meter walk, and chair stands, which predicts disability and mortality in older adults and cancer patients. Each of the 3 tests are scored from 0-4 and summed for a total scale range of 0-12, with higher scores indicating better physical function.
Short Physical Performance Battery Score at 6 months follow-up | at 6 months follow-up
  Physical performance at 6 months follow-up, measured by the Short Physical Performance Battery (SPPB), a 10-minute provider-administered test of balance, 4-meter walk, and chair stands, which predicts disability and mortality in older adults and cancer patients. Each of the 3 tests are scored from 0-4 and summed for a total scale range of 0-12, with higher scores indicating better physical function.
Patient-Reported Outcomes Version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) Score at Post-RT | at end of RT, average of 10 days
  Patient reported toxicity outcomes as measured using the PRO-CTCAE scale at post-RT. The PRO-CTCAE is a 5-minute survey, integrating patient perspectives into clinicians' reporting of treatment toxicity. It is validated for use in medical and radiation oncology and has revealed clinician underreporting of toxicity severity in older patients. The survey is scored on a 0-5-point scale, where higher outcomes indicate worse health outcomes.
PRO-CTCAE Score at 1 month follow-up | at 1 month follow-up
  Patient reported toxicity outcomes as measured using the PRO-CTCAE scale at 1 month follow-up. The PRO-CTCAE is a 5-minute survey, integrating patient perspectives into clinicians' reporting of treatment toxicity. It is validated for use in medical and radiation oncology and has revealed clinician underreporting of toxicity severity in older patients. The survey is scored on a 0-5-point scale, where higher outcomes indicate worse health outcomes.
PRO-CTCAE Score at 3 months follow-up | at 3 months follow-up
  Patient reported toxicity outcomes as measured using the PRO-CTCAE scale at 3 months follow-up. The PRO-CTCAE is a 5-minute survey, integrating patient perspectives into clinicians' reporting of treatment toxicity. It is validated for use in medical and radiation oncology and has revealed clinician underreporting of toxicity severity in older patients. The survey is scored on a 0-5-point scale, where higher outcomes indicate worse health outcomes.
PRO-CTCAE Score at 6 months follow-up | at 6 months follow-up
  Patient reported toxicity outcomes as measured using the PRO-CTCAE scale at 6 months follow-up. The PRO-CTCAE is a 5-minute survey, integrating patient perspectives into clinicians' reporting of treatment toxicity. It is validated for use in medical and radiation oncology and has revealed clinician underreporting of toxicity severity in older patients. The survey is scored on a 0-5-point scale, where higher outcomes indicate worse health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Dharmarajan, MD, MSc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- One Gustave L Levy Place, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD data.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT05721053/ICF_000.pdf